CLINICAL TRIAL: NCT03147287
Title: Palbociclib After CDK and Endocrine Therapy (PACE): A Randomized Phase II Study of Fulvestrant, Palbociclib, and Avelumab for Endocrine Pre-treated ER+/HER2- Metastatic Breast Cancer
Brief Title: Palbociclib After CDK and Endocrine Therapy (PACE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Senior Physician, Susan F Smith Center for Women's Cancers, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-101
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fulvestrant (Active Comparator): -Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly
  Interventions: Drug: Fulvestrant
- Fulvestrant with Palbociclib (Experimental): -Palbociclib should be taken orally, once per day for 21 days on a 28 days cyclye -Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly
  Interventions: Drug: Palbociclib; Drug: Fulvestrant
- Fulvestrant with Palbociclib and Avelumab (Experimental): -Palbociclib should be taken orally, once per day for 21 days on a 28 days cyclye -Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly -Avelumab will be administered intravebously once every 2 weeks
  Interventions: Drug: Palbociclib; Drug: Fulvestrant; Drug: Avelumab

INTERVENTIONS:
Drug: Palbociclib — Palbociclib is a drug that may stop cancer cells from growing
  Other Names: Ibrance
  Arms: Fulvestrant with Palbociclib; Fulvestrant with Palbociclib and Avelumab
Drug: Fulvestrant — Fulvestrant prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen
  Other Names: Faslodex
Drug: Avelumab — Avelumab is an antibody designed to block the PD-1 pathway and helps the immune system in detecting and fighting cancer cells
  Other Names: Bavencio
  Arms: Fulvestrant with Palbociclib and Avelumab

SUMMARY:
This research study is studying three combinations of drugs as treatments for breast cancer. The drugs involved in this study are: -Fulvestrant -Fulvestrant with Palbociclib -Fulvestrant with Palbociclib and Avelumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied and the researchers are trying to find out more about it- for example, the side effects it may cause, and the activity of a drug, or combination of drugs, against a cancer. In this research study, the investigators are evaluating the activity of fulvestrant alone, fulvestrant and palbociclib, or fulvestrant, palbociclib, and avelumab combined, in participants with metastatic hormone receptor positive HER2 negative breast cancer that has previously stopped responding to prior palbociclib and endocrine therapy. The FDA (the U.S. Food and Drug Administration) has approved both palbociclib and fulvestrant as treatment options for this disease, however the use of palbociclib has not been studied in people who have previously been treated with palbociclib. The FDA has not approved avelumab as a treatment for any disease. Palbociclib is a drug that may stop cancer cells from growing. Palbociclib blocks activity of two closely related enzymes (proteins that help chemical reactions in the body occur), called Cyclin Dependent Kinases 4 and 6 (CDK 4/6). These proteins are part of a pathway, or a sequence of steps, which is known to promote cancer cell growth. Laboratory testing has shown that palbociclib may stop the growth of hormone receptor positive breast cancer. Palbociclib is FDA-approved as therapy for metastatic hormone receptor positive HER2 negative breast cancer in combination with endocrine therapy in the first line setting, and in combination with fulvestrant for pre-treated disease. It is not known whether cancers that have grown despite prior palbociclib treatment are still sensitive to palbociclib. Endocrine therapy prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen. During this study, the endocrine therapy will be fulvestrant. Fulvestrant is a drug that is approved by the FDA for treatment of metastatic hormone receptor positive breast cancer. The immune system is the body's natural defense against disease. The immune system sends a type of cells called T cells throughout the body to detect and fight infections and diseases-including cancers. One way the immune system controls the activity of T cells is through the PD-1 (programmed cell death protein-1) pathway. However, some cancer cells hide from T-cell attack by taking control of the PD-1 pathway and this stops T cells from attacking cancer cells. Avelumab is an antibody designed to block the PD-1 pathway and helps the immune system in detecting and fighting cancer cells. An antibody is a protein produced by the body's immune system when it detects harmful substances. Previous studies show that the administration of antibodies which block the PD-1 pathway can lead to tumor destruction. In the laboratory, adding avelumab to fulvestrant and palbociclib appears to improve effectiveness. It is not known whether this is true in humans

ELIGIBILITY:
Inclusion Criteria: -Participants must have histologically confirmed hormone receptor positive (HR+) HER2 negative metastatic or locally recurrent unresectable invasive breast cancer. ER, PR and HER2 measurements should be performed according to institutional guidelines, in a CLIA-approved setting. Cut-off values for positive/negative staining should be in accordance with current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines. -Men and pre- and postmenopausal women are eligible. Ongoing monthly GNRH agonist is required in pre-menopausal women or male participants for at least 4 weeks prior to study entry. -Participants must have radiological or objective evidence of progression on an endocrine and CDK 4/6 inhibitor regimen in the metastatic setting, and/or relapse/progression during or within 12 months of completion of an endocrine and CDK4/6 inhibitor regimen in the adjuvant setting. --Participants must have previously been exposed to CDK4/6 inhibitor therapy in combination with endocrine therapy. Exposure to any prior CDK4/6 inhibitor, (including palbociclib, abemaciclib, and ribociclib) is allowed. Patients may have a line of endocrine therapy after combination endocrine and CDK4/6 inhibitor exposure. --Participants must have remained on prior endocrine and CDK4/6 therapy in the metastatic setting without progression for at least 6 months prior to study entry. --It is not mandatory to have a CDK 4/6 inhibitor containing regimen as the most recent treatment. -Participants may have 0-1 prior lines of cytotoxic chemotherapy in the metastatic setting. -Prior endocrine therapy in the metastatic setting may include any aromatase inhibitor (AI) or tamoxifen, but may not include prior fulvestrant. In the metastatic setting, 1-2 prior lines of endocrine therapy are allowed. -Participants may have received radiotherapy for palliative purpose, but must not be experiencing > grade 1 treatment related toxicities, and must have completed treatment > 14 days prior to registration. -Age ≥18 years. Because no dosing or adverse event data are currently available on the use of study agents in participants <18 years of age, children are excluded from this study. -ECOG performance status 0-1 (see Appendix A). -Participants must have normal organ and marrow function as defined below: -Absolute neutrophil count > 1,500/µL --Platelets > 100,000/µL --Hemoglobin > 9g/dL --Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (participants with documented Gilbert's disease are allowed total bilirubin up to 1.5X ULN) --AST (SGOT)/ALT (SGPT) < 2.5 x institutional ULN, or ≤ 5 x ULN for subjects with documented metastatic disease to the liver. --Creatinine < institutional ULN or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional ULN. --Baseline QTc < 480 ms -The effects of palbociclib and avelumab on the developing human fetus are unknown. If, for any reason, a woman should become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately. Women of childbearing age, women who are made postmenopausal through use of GNRH agonists, and men must agree to use adequate contraception for the duration of protocol treatment and for at least 60 days after the last dose of study medication if the risk of contraception exists. -Adequate contraception is defined as one highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the participant and/or partner. -Highly Effective Non-Hormonal Contraception -Methods of birth control which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly are considered highly-effective forms of contraception. -The following non-hormonal methods of contraception are acceptable: --True abstinence when this is in line with the preferred and usual lifestyle of the participant. [Periodic abstinence (e.g., calendar, ovulation, symptothermal post-ovulation methods) and withdrawal are not acceptable methods of contraception]. --Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female participants, the vasectomized male partner should be the sole partner. OR -Effective Non-Hormonal Contraception Alternatively two of the following effective forms of contraception may be used instead: --Placement of non-hormonal intrauterine device (IUD) or intrauterine system (IUS). Consideration should be given to the type of device being used, as there is higher failure rates quoted for certain types, e.g., steel or copper wire. --Condom with spermicidal foam/gel/film/cream/suppository. --Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. --The use of barrier contraceptives should always be supplemented with the use of spermicide. The following should be noted: --Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore, the use of additional spermicides does confer additional theoretical contraceptive protection. --However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone. It should be noted that two forms of effective contraception are required. A double barrier method is acceptable, which is defined as condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream /suppository. -Premenopausal women must have a negative serum or urine pregnancy test. Pregnancy testing does not need to be pursued in female participants who are: --Age > 60 years; or --Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more AND estrogen (estradiol) levels within postmenopausal range; or --Status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation. -Participant must be able to swallow and retain oral medication. -Ability to understand and the willingness to sign a written informed consent document Exclusion Criteria: -Participants who have had endocrine, chemotherapy, and/or biologic therapy within 14 days prior to entering the study or those who have not recovered from any prior treatment-related toxicities (must recover to no more than grade 1. Alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 toxicity not constituting a safety risk based on investigator's judgment are acceptable). -Participants who are receiving concurrent therapy with other investigational agents. -Rapidly progressive, symptomatic, visceral spread of disease placing participant at risk of life-threatening complications in the short term. -Participants with active brain metastases. Stable treated brain metastases are allowed (this includes participants who have documented radiologic stability at least 4 weeks after radiotherapy, and do not require systemic steroids for management of symptoms from CNS metastatic lesions). -Participants who have discontinued prior palbociclib for toxicity, or have needed more than one dose or schedule reduction for toxicity from prior palbociclib therapy. If a participant required a single dose reduction during prior palbociclib therapy and tolerated it well, for example prior dosing at 100 mg qd 3 weeks on 1 week off schedule, than that dose may be selected for this trial. -History of allergic reactions to palbociclib or attributed to compounds of similar chemical or biologic composition to palbociclib. -Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3) -Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A isoenzymes are ineligible. Lists including medications and substances known or with the potential to interact with the CYP3A isoenzymes are provided in Appendix B, and can also be found within Section 5.4. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product. -Current use of drugs listed in Appendix C that are known to prolong the QT interval (See Appendix C) -Prior organ transplantation including allogenic stem-cell transplantation -Current use of immunosuppressive medication, except for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication). -Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring systemic therapy, clinically significant cardiovascular disease including: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication, uncontrolled diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation. -Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Participants with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. -Known history of testing positive for HIV or known acquired immunodeficiency syndrome, or need to receive combination antiretroviral therapy for HIV -Known history of immune-mediated conditions including colitis, inflammatory bowel disease requiring steroid or immunosuppressive therapy, pneumonitis, or pulmonary fibrosis. -Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive) -Live vaccination within 4 weeks of the first dose of avelumab -Pregnant women are excluded from this study because effect of palbociclib and avelumab on a developing fetus is unknown. Breastfeeding should be discontinued prior to entry onto the study. -Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Erica L Mayer, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (22):
- United States (22):
  - University of Miami, Miami, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - The University of Kansas Cancer Center - North, Kansas City, Kansas
  - The University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at St. Elizabeth's Medical Center, Brighton, Massachusetts
  - DF/BWCC at Milford Regional Medical Center, Milford, Massachusetts
  - DF/BWCC in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - The University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University, St Louis, Missouri
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University, Houston, Texas
  - Aurora Cancer Care, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer EL, Ren Y, Wagle N, Mahtani R, Ma C, DeMichele A, Cristofanilli M, Meisel J, Miller KD, Abdou Y, Riley EC, Qamar R, Sharma P, Reid S, Sinclair N, Faggen M, Block CC, Ko N, Partridge AH, Chen WY, DeMeo M, Attaya V, Okpoebo A, Alberti J, Liu Y, Gauthier E, Burstein HJ, Regan MM, Tolaney SM. PACE: A Randomized Phase II Study of Fulvestrant, Palbociclib, and Avelumab After Progression on Cyclin-Dependent Kinase 4/6 Inhibitor and Aromatase Inhibitor for Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor-Negative Metastatic Breast Cancer. J Clin Oncol. 2024 Jun 10;42(17):2050-2060. doi: 10.1200/JCO.23.01940. Epub 2024 Mar 21. PMID 38513188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 sites that randomized 220 participants between September 5, 2017 and February 23 2022. Eligible participants were to have HR+/HER2- advanced breast cancer, with prior objective progression on an endocrine + CDK4/6 inhibitor regimen; 0-1 prior lines of chemotherapy for ABC, no prior fulvestrant.
Groups:
- Fulvestrant With Palbociclib: * Palbociclib should be taken orally, once per day for 21 days on a 28 days cyclye
  * Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly
  Palbociclib: Palbociclib is a drug that may stop cancer cells from growing
  Fulvestrant: Fulvestrant prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen
- Fulvestrant With Palbociclib and Avelumab: * Palbociclib should be taken orally, once per day for 21 days on a 28 days cyclye
  * Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly
  * Avelumab will be administered intravebously once every 2 weeks
  Palbociclib: Palbociclib is a drug that may stop cancer cells from growing
  Fulvestrant: Fulvestrant prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen
  Avelumab: Avelumab is an antibody designed to block the PD-1 pathway and helps the immune system in detecting and fighting cancer cells
Period: Overall Study
Arm/Group | Fulvestrant | Fulvestrant With Palbociclib | Fulvestrant With Palbociclib and Avelumab
Started | 55 | 111 | 54
Completed | 0 | 0 | 0
Not Completed | 55 | 111 | 54
Not completed — Randomized Not Treated | 2 | 1 | 1
Not completed — Progressive Disease RECIST | 31 | 72 | 32
Not completed — Progressive Disease not RECIST | 13 | 21 | 13
Not completed — Physician Decision | 1 | 2 | 1
Not completed — Intercurrent illness | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Patient Non-Compliance | 0 | 2 | 0
Not completed — Patient moved | 0 | 1 | 0
Not completed — Arm A crossover without PD | 1 | 0 | 0
Not completed — Ongoing at date of cut-off (11 Jul 2022) | 5 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Fulvestrant: -Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly Fulvestrant: Fulvestrant prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen
- Fulvestrant With Palbociclib: -Palbociclib should be taken orally, once per day for 21 days on a 28 days cyclye -Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly Palbociclib: Palbociclib is a drug that may stop cancer cells from growing Fulvestrant: Fulvestrant prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen
- Fulvestrant With Palbociclib and Avelumab: -Palbociclib should be taken orally, once per day for 21 days on a 28 days cyclye -Fulvestrant will be administered in the clinic as two IM injections on Cycle 1 Days 1, 15, then monthly -Avelumab will be administered intravebously once every 2 weeks Palbociclib: Palbociclib is a drug that may stop cancer cells from growing Fulvestrant: Fulvestrant prevents growth of hormone receptor positive breast cancer by blocking stimulation of cancer cells by estrogen Avelumab: Avelumab is an antibody designed to block the PD-1 pathway and helps the immune system in detecting and fighting cancer cells
- Total: Total of all reporting groups
Arm/Group | Fulvestrant | Fulvestrant With Palbociclib | Fulvestrant With Palbociclib and Avelumab | Total
Number analyzed (Participants) | 55 | 111 | 54 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.2) | 54.2 (11.9) | 57.0 (11.4) | 55.9 (11.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex and menopausal status: Male | 0 | 2 | 0 | 2
  Sex and menopausal status: Female premenopausal | 8 | 22 | 10 | 40
  Sex and menopausal status: Female postmenopausal | 47 | 87 | 44 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 47 | 88 | 44 | 179
  Race: Black or African American | 3 | 13 | 4 | 20
  Race: Asian | 0 | 4 | 3 | 7
  Race: More Than One Race | 0 | 2 | 1 | 3
  Race: Other | 5 | 4 | 2 | 11
Prior chemotherapy between prior CDK4/6i and randomization (stratification factor) [Count of Participants; unit: Participants] | 3 | 4 | 2 | 9
De novo metastatic breast cancer [Count of Participants; unit: Participants] | 28 | 40 | 20 | 88
Visceral disease [Count of Participants; unit: Participants] | 29 | 70 | 33 | 132

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), According to RECIST v1.1 Criteria (Investigator Assessment)
Description: Progression-Free Survival (PFS), according to RECIST v1.1 criteria (investigator assessment): the time from randomization to the earlier of progression or death due to any cause. Participants alive without disease progression were censored at date of last disease assessment (tumor assessments). The date of progression was the first date that recurrent or progressive disease was objectively documented; if death was the defining event, it must have happened within 2 intervals of the last disease assessment, otherwise PFS was censored at last disease assessment. The length of PFS was calculated as PFS time (months) =[progression/death date(censor date) - randomization date + 1]/30.4375.
Time Frame: Tumor were assessed every 8 weeks until 24 weeks, then every 12 weeks. The median PFS follow-up time at database lock was 12.1 months (range 1 day to 50.1 months).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Fulvestrant | Fulvestrant With Palbociclib | Fulvestrant With Palbociclib and Avelumab
Number analyzed (Participants) | 55 | 111 | 54
months | 4.8 [2.1 to 8.2] | 4.6 [3.6 to 5.9] | 8.1 [3.2 to 10.7]
Statistical Analysis 1: Comparison: Fulvestrant vs Fulvestrant With Palbociclib; The primary objective was investigated by comparing the PFS distributions between two treatment arms using a logrank test with one-sided α level of 0.05 (H0: PFS1≤PFS2; HA: PFS1>PFS2). Hazard ratios were estimated from a Cox PH model (F+P / F, so that HR<1 indicates reduced hazard of PFS event with F+P), with two sided 90% CIs (Wald) to align with the design and testing; Test type: Superiority; p = 0.62, Log Rank — We reported two-sided p-values corresponding to two-sided α level of 0.10. The test statistic and p-value were taken from the Cox proportional hazards model score test; The SAP intended stratified tests and models, however one stratum was only 9 patients making implementation of stratification questionable; Hazard Ratio (HR) = 1.11, 90% CI 2-sided [0.79 to 1.55] — We checked the proportional hazards assumption by visually assessing the plot of log( log(survival)) vs log of survival times according to treatment assignment for parallelism. This was done overall and according to stratum

2. Secondary Outcome: Overall Response Rate, According to RECIST v1.1 Criteria (Investigator Assessment)
Description: Objective Response (OR): best overall response of complete response or partial response. Response was primarily evaluated in this study using the criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). For example, target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. See RECIST 1.1 manuscript for further details on overall assessment based on target lesions, non-target lesions and new lesions. The Overall Response Rate (with 2-sided 90% CIs) were estimated according to treatment assignment and subgroup.
Time Frame: Tumor were assessed every 8 weeks until 24 weeks, then every 12 weeks. The median follow-up time for overall response rate at database lock was 12.1 months (range 1 day to 50.1 months).
Measure: Number (90% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Fulvestrant | Fulvestrant With Palbociclib | Fulvestrant With Palbociclib and Avelumab
Number analyzed (Participants) | 55 | 111 | 54
percentage of participants analyzed | 7.3 [1.5 to 13.0] | 9.0 [4.5 to 13.5] | 13.0 [5.4 to 20.5]
Statistical Analysis 1: Comparison: Fulvestrant vs Fulvestrant With Palbociclib; The objective response was reported with two-sided 90% CI and compared between two treatment arms using a (unstratified) Fisher's exact test;; Test type: Superiority; p = 1.000, Fisher Exact — P-value is two sided, for hypothesis test with two-sided α=0.10

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability)
Description: The frequency (and %) of patients who are reported as having grade 3-5 treatment-related adverse events were summarized. From starting the first dose of study treatment to 30 days (90 days for arm C) after last dose administration of study treatment or study discontinuation, whichever was earlier. Afterwards only SAEs attributed to study treatment were reported.
Time Frame: The median follow-up time for adverse event was 5.4 months (range 1.6 months to 51.2 months).
Population: Of 220 patients in the ITT population, 216 initiated protocol-assigned treatment(s) and comprise the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant | Fulvestrant With Palbociclib | Fulvestrant With Palbociclib and Avelumab
Number analyzed (Participants) | 53 | 110 | 53
Participants | 1 | 46 | 37

ADVERSE EVENTS:
Time Frame: After starting the first dose of study treatment and ended 30 days (90 days for arm C) after last dose administration of study treatment or study discontinuation/termination, whichever was earlier. Afterwards only SAEs attributed to study treatment were reported. The median follow-up time for adverse events was 5.4 months (range 1.6 months to 51.2 months). The median follow-up time for all-cause mortality was 23.6 months (range 1 day to 50.2 months).
Description: The maximum grade of each adverse event (AE) type was summarized as frequency (and %) of patients experiencing the AE, tabulated according to body system and AE type, separately according to treatment group. Serious Adverse Events (SAEs) were defined as treatment-related grade 3-5 adverse events. Other Adverse Events (OAEs) were defined as adverse events that are not SAEs. All 220 patients were assessed for mortality, and the 216 patients who initiated study treatment were assessed for AEs.
Arm/Group | Fulvestrant | Fulvestrant With Palbociclib | Fulvestrant With Palbociclib and Avelumab
All-Cause Mortality (participants affected / at risk) | 23/55 | 43/111 | 17/54
Serious Adverse Events (participants affected / at risk) | 1/53 | 46/110 | 37/53
Other Adverse Events (participants affected / at risk) | 47/53 | 105/110 | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant (N=53) | Fulvestrant With Palbociclib (N=110) | Fulvestrant With Palbociclib and Avelumab (N=53)
Anemia (Blood and lymphatic system disorders) | 0 | 5 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1
Infustion related reaction (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 3
Irritability (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Cardiac troponin T increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 4 | 6
Neutrophil count decreased (Investigations) | 0 | 36 | 26
Platelet count decreased (Investigations) | 0 | 1 | 2
White blood cell decreased (Investigations) | 0 | 15 | 11
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant (N=53) | Fulvestrant With Palbociclib (N=110) | Fulvestrant With Palbociclib and Avelumab (N=53)
Anemia (Blood and lymphatic system disorders) | 8 | 25 | 21
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 2
Hypothyroidism (Endocrine disorders) | 2 | 1 | 4
Blurred vision (Eye disorders) | 1 | 3 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 2 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 2
Eye pain (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Papilledema (Eye disorders) | 1 | 0 | 0
Scleral disorder (Eye disorders) | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 6
Ascites (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 15 | 14
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 21 | 14
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 3 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 13 | 8
Nausea (Gastrointestinal disorders) | 8 | 20 | 14
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 4 | 6 | 4
Infusion related reaction (General disorders) | 1 | 1 | 4
Chills (General disorders) | 1 | 2 | 5
Edema limbs (General disorders) | 0 | 9 | 3
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 23 | 46 | 44
Fever (General disorders) | 1 | 4 | 9
Flu like symptoms (General disorders) | 0 | 3 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 1 | 4
Injection site reaction (General disorders) | 6 | 13 | 3
Irritability (General disorders) | 1 | 0 | 1
Localized edema (General disorders) | 1 | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 3 | 2
Pain (General disorders) | 8 | 20 | 13
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 4 | 3 | 3
Laryngitis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 3
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 2 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0
Skin infection (Infections and infestations) | 0 | 4 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2 | 4
Urinary tract infection (Infections and infestations) | 1 | 3 | 5
Uterine infection (Infections and infestations) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fallopian tube anastomotic leak (Injury, poisoning and procedural complications) | 0 | 3 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 3 | 0
Intraoperative hepatobiliary injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 1 | 5
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 0 | 0
Uterine anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 8 | 10 | 7
Alkaline phosphatase increased (Investigations) | 8 | 14 | 2
Aspartate aminotransferase increased (Investigations) | 12 | 14 | 10
Blood bilirubin increased (Investigations) | 1 | 4 | 3
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0
CPK increased (Investigations) | 1 | 1 | 5
Cardiac troponin I increased (Investigations) | 0 | 1 | 1
Creatinine increased (Investigations) | 0 | 8 | 10
INR increased (Investigations) | 0 | 1 | 0
Investigations - Other, specify (Investigations) | 1 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 7 | 21 | 13
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 59 | 35
Platelet count decreased (Investigations) | 2 | 17 | 16
Weight gain (Investigations) | 1 | 1 | 2
Weight loss (Investigations) | 0 | 3 | 6
White blood cell decreased (Investigations) | 7 | 37 | 22
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 9 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 13 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 7 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 7 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 4 | 7
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 17 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 10 | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Growth suppression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6 | 14
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Brachial plexopathy (Nervous system disorders) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 2 | 1
Concentration impairment (Nervous system disorders) | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 2 | 5 | 1
Dizziness (Nervous system disorders) | 4 | 7 | 10
Dysesthesia (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 4
Edema cerebral (Nervous system disorders) | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 9 | 14 | 7
Memory impairment (Nervous system disorders) | 1 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 4 | 4
Presyncope (Nervous system disorders) | 1 | 0 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 4 | 4
Confusion (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 4 | 5 | 2
Insomnia (Psychiatric disorders) | 4 | 15 | 10
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 2
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 5
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 2 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 15 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 3 | 18 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 8 | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 8 | 5
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 | 3 | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 1
Hot flashes (Vascular disorders) | 10 | 6 | 3
Hypertension (Vascular disorders) | 7 | 16 | 7
Hypotension (Vascular disorders) | 3 | 1 | 1
Lymphedema (Vascular disorders) | 1 | 5 | 0
Thromboembolic event (Vascular disorders) | 0 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03147287/Prot_SAP_000.pdf